CLINICAL TRIAL: NCT04563611
Title: Effect of Turkish Get Up and Hamstring Exercises on Hamstring Muscle Function, Injury Risk, Agility and Cognitive Function
Brief Title: Effect of Exercises on Hamstring Muscle Function, Injury Risk, Agility and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, caglar soylu, Çağlar Soylu, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-79/38
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Hamstring Muscles; Muscle Function; Cognitive Function; Turkish Get Up
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Healthy recreational people aged between 18-25 will assign to this study. The participants will randomly be allocated four groups (Nordic protocol group, Supine sliding leg curls group, Turkish Get Up (TGU) and control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Muscle strength (No Intervention): Participants hamstring muscle strengths will be evaluated with ISOMED 2000 isokinetic dynamometer
- Hamstring Flexibility (No Intervention): In this study, Individuals' evaluations of hamstring flexibility will be assessed by the active knee extension test (ICC: 0.96) with maximum hip flexion.
- Cognitive Function (No Intervention): The lower (reaction time and visual-perceptual ability) and upper level (working memory, inhibitory control, and cognitive flexibility) cognitive functions of the individuals participating in the study will be evaluated with the computer assisted CNSVS test battery
- Injury risk (No Intervention): Injury risk analysis of individuals will be made using the strength differences between the two sides, H: Q ratios (conventional and functional ratio) and functional movement screen (FMS), which will be obtained from the isokinetic measurement results.
- Nordic hamstring exercise (Experimental): To perform this exercise, participants will be asked to stand in an upright position on their knees. The hands and arms will be positioned on the chest and held by the physical therapist at the heels of the individuals. The individual will then be asked to lower the upper body forward as slowly as possible. Verbal commands will be given throughout the movement so that the hip and trunk smoothness is not disturbed
  Interventions: Other: Nordic hamstring exercise; Other: Control Group
- Supine Sliding Leg Curls (Experimental): The persons will be started to exercise in the hook position, with hands-on their back, with their knees next to the body, in a flexion position of approximately 60 °. Participants will be asked to first build a bridge, then maintain this position and slowly slide the slippery apparatus under their feet to bring their knees to full extension.
  Interventions: Other: Askling L-Protocol; Other: Control Group
- Turkish Get-up exercise (Experimental): TG exercise, in 7 different steps (1. Starting position, 2. Supine girya lifting, 3. Elbow supported kettlebell lifting, 4. Hand supported kettlebell lifting, 5. High bridge, 6. Half above knee and lunge position, 7. Standing up) and the return of these different steps.
  Interventions: Other: Turkish Get-up exercise; Other: Control Group
- Agility (No Intervention): Agility performances of individuals will be evaluated with the Agility T-test.

INTERVENTIONS:
Other: Turkish Get-up exercise — TG exercise, in 7 different steps (1. Starting position, 2. Supine girya lifting, 3. Elbow supported kettlebell lifting, 4. Hand supported kettlebell lifting, 5. High bridge, 6. Half above knee and lunge position, 7. Standing up) and the return of these different steps.
  Arms: Turkish Get-up exercise
Other: Askling L-Protocol — he protocol consists of 3 different exercises. These are exercise 1 aimed at increasing flexibility, exercise 2 providing strength and trunk / pelvis stabilization, and exercise 3 aiming at specific strengthening. Pain is not allowed to be provoked when performing the exercises.
  Arms: Supine Sliding Leg Curls
Other: Nordic hamstring exercise — To perform this exercise, participants will be asked to stand in an upright position on their knees. Hands and arms will be positioned on the chest and the individuals will be held by the physiotherapist at their heels. The individual will then be asked to lower the upper body forward as slowly as possible. Verbal commands will be given throughout the movement so that the hip and trunk smoothness is not disturbed.
  Arms: Nordic hamstring exercise
Other: Control Group — No exercise will be applied to the individuals in the control group. At the end of the 6-week period, all parameters will be evaluated again.
  Arms: Nordic hamstring exercise; Supine Sliding Leg Curls; Turkish Get-up exercise

SUMMARY:
Hamstring muscle injuries (HMI) occurs frequently during excessive motions of the physiologic capability of these muscles. It is reported in the literature that impairments in muscle architecture, such as a decrease in the eccentric strength of the hamstring muscles of the knee (lengthening and contraction of the muscle), delay in the reaction time of the hamstring muscles, overactivity of the hamstring muscles, a decrease in the length of the hamstring muscle fibers, and inadequate cognitive functions may lead to HMI. Preventive and therapeutic exercises of HMI consist many different eccentric exercises, such as the Askling L-protocol and particularly Nordic hamstring exercise, for increasing the hamstring flexibility. However, it has been stated in recent studies that hamstring muscles should not be focused on alone, and a holistic exercise intervention that includes and addresses the present risk factors related to HMI is needed. Within our knowledge, the effect of a defined or improved holistic exercise approach to prevent and/or treat HMI has not been studied in the literature. Considering the risk factors underlying HMI, an exercise involving a holistic approach is needed to prevent all the risk factors. Turkish Get Up (TGU) exercise is a kind of cognitive exercise which activates all muscles and let to contract simultaneously during standing up from the supine position and turning back in 7 stages. Since the exercise originates from former Turkish athletes, it has been included in the literature as TGU. Hence, the exercise originates from former Turkish athletes, it has called as TGU. TGU exercise improves the effective and strong transition ability of the body while developing the pattern of standing up from the lying position on the floor and turning back by increasing condition/ endurance. Meanwhile, this exercise is a progressive coordinative and cognitive exercise, it requires completing each step before the next movement.

The role of cognitive skills and neuroscience in the interpretation, prediction and improvement of sports performance is getting popular in recent years. Previous researches reported that athletes with reduced cognitive skills had lower sportive achievements. It has also stated that the impairment in cognitive skills tend muscles to be injured. However, no studies that investigate the effectiveness of cognitive function in preventing HMI have been encountered. So, the present study will be the first study investigating effects of a special exercise addressing cognitive function which is generally ignored in the treatment of HMI.

It is aimed to figure out whether Turkish Get Up exercise or Supine sliding leg curls and Nordic Hamstring exercises are more effective on hamstring muscle function, ınjury risk, agility and cognitive function.

Healthy recreational people aged between 18-25 will assign to this study. The participants will randomly be allocated four groups (Nordic protocol group, Supine sliding leg curls group, Turkish Get Up (TGU) and control group). The exercise protocols will be applied two days a week for 6 weeks, and the control group will receive no special exercise training. Participants' hamstring muscle strengths will be evaluated with ISOMED 2000 isokinetic dynamometer, the hamstring flexibility with digital inclinometer device, injury risk with FMS™, agility with T-agility test, and the cognitive function with CNS Vital Signs in computer environment at baseline and 6 weeks after interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18-25
2. Body mass index (BMI) being between 18.5-24.9 kg / m 2
3. Volunteering to participate in the study
4. Having the skills to do the tests and exercises to be applied
5. Being a healthy recreationally active male individual (Individuals with sufficient physical activity level according to the International Physical Activity Questionnaire (IPAQ) Short form (> 3000 metabolic equivalent (MET) -min / week) will be included)

Exclusion Criteria:

1. Having a history of lower extremity injury and / or hamstring strain within the past year
2. Having a sensory problem that prevents participation in the study
3. Have any musculoskeletal, neurological, respiratory, or cardiovascular risk factors that limit exercise
4. Using drugs or nutritional supplements that can be considered doping according to the World Anti-Doping Agency (WADA)
5. Having a history of malignant disease

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Hamstring Muscle Strength | 6 weeks
  Participants hamstring muscle strengths will be evaluated with ISOMED 2000 isokinetic dynamometer
Hamstring Flexibility | 6 weeks
  In this study, Individuals' evaluations of hamstring flexibility will be assessed by the active knee extension test (ICC: 0.96) with maximum hip flexion.
Cognitive Function | 6 weeks
  The lower (reaction time and visual-perceptual ability) and upper level (working memory, inhibitory control, and cognitive flexibility) cognitive functions of the individuals participating in the study will be evaluated with the computer assisted CNSVS test battery
Injury risk | 6 weeks
  Injury risk analysis of individuals will be made using the strength differences between the two sides, H: Q ratios (conventional and functional ratio) and functional movement screen (FMS), which will be obtained from the isokinetic measurement results.
Agility | 6 weeks
  Agility performances of individuals will be evaluated with the Agility T test.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No